CLINICAL TRIAL: NCT04321941
Title: Randomised, Open, Non-inferiority Within Patient-controlled Trial Evaluating the Diagnostic Usefulness of Lumentin® 44 When Used as Contrast Agent in CT-enterography as Compared to MRI- Enterography in Patients With Small Bowel Crohn's Disease
Brief Title: Trial Evaluating the Diagnostic Usefulness of Lumentin® 44 When Used as Contrast Agent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lument AB (Industry)
Collaborators: LINK Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: LUM-002; 2019-002093-32 (EudraCT Number)
Record Dates: First submitted 2020-03-24; First posted 2020-03-25 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Within patient comparison of diagnostic methods
Who Masked: Outcomes Assessor
Masking Description: Blinded evaluation of MRE and CTE images respectively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTE (Computerised Tomography Enterography) (Experimental): CTE examination performed with experimental contrast agent, Lumentin.
  Interventions: Diagnostic Test: Lumentin
- MRE (Magnetic Resonance Enterography) (Active Comparator): Comparative diagnostic method performed with the contrast agent Movprep®
  Interventions: Diagnostic Test: Movprep

INTERVENTIONS:
Diagnostic Test: Lumentin — Contrast agent used in combination with CTE
  Arms: CTE (Computerised Tomography Enterography)
Diagnostic Test: Movprep — Contrast agent used in combination with MRE
  Arms: MRE (Magnetic Resonance Enterography)

SUMMARY:
The trial is a phase 2 randomised, open, non-inferiority within patient-controlled multi-centre trial.

Male and female subjects with a diagnosis of Crohn´s Disease and a clinical indication for an MRE examination, who are at least 18 years of age and who provide a written informed consent, will be eligible for inclusion.

The trial period will be up to 16 weeks and consists of 7 visits (see schedule of events). All patients who have attended at least 1 of the Magnetic Resonance Enterography (MRE)/Computerised Tomography Enterography (CTE) examinations should go through the end of treatment procedures at visit 7.

Subjects will attend two examinations during the course of the trial:

* A CTE
* An MRE The Crohn's disease activity will be assessed radiologically on the MRE and CTE scans by identifying the presence and severity of a number of morphologic entities and dynamic signs in the SB and colon as described in the RCDAS.

Additional evaluation of CD activity and disease complication on the MRE and CTE images will be performed using the CDMRIS scale and Lémann Index respectively

DETAILED DESCRIPTION:
The trial is a phase 2 randomised, open, non-inferiority within patient-controlled multi-centre trial.

Patient recruitment will take place at 1 or more study centres by clinicians specialised in gastroenterology. MRE and CTE examinations will be performed at the department of Radiology at a hospital or private practise that performs radiology. Participating radiology department or private practice need to be certified to perform the examination at Skåne University Hospital, SUS, Malmö, Sweden.

Male and female subjects with a diagnosis of CD and a clinical indication for an MRE examination, who are at least 18 years of age and who provide a written informed consent, will be eligible for inclusion.

The trial period will be up to 16 weeks and consists of 7 visits (see schedule of events). All patients who have attended at least 1 of the MRE/CTE examinations should go through the end of treatment procedures at visit 7.

Subjects interested in participating in the trial will be screened for eligibility at visit 1. After receiving information about the trial according to the procedures for subject information and consent (see section 14.3) and found eligible according to the in-/exclusion criteria, patients will be included in the trial and randomised. After randomisation, the subject's demography, medical history and concomitant illness and medical treatment will be noted

Subjects will attend two examinations during the course of the trial:

* A CTE
* An MRE The order in which the MRE and CTE-L is performed will be randomised. Date and time for the patient's MRE examination will be booked at the department of radiology when the subject have been randomised. The date of CTE examination will then be booked two to three weeks apart from the MRE, either before or after according to the randomisation, to ensure both a proper washout period of given medical compounds and a minimal risk of change in status of the disease.

The Crohn's disease activity will be assessed radiologically on the MRE and CTE scans by identifying the presence and severity of a number of morphologic entities and dynamic signs in the SB and colon as described in the RCDAS.

The radiologist assessment, according to the RCDAS, of the CTE and MRE examinations will be performed by the investigators specialised in abdominal imaging at the department of radiology. The radiologist assessment of one patient's CTE and MRE examinations will not be performed by the same investigator in order to avoid that one assessment influence the other. Appointment of assessor for each examination will be performed by randomisation.

Pseudonymised assessment of CTE and MRE scans will be performed in batches of approximately 5 scans. Patient identification details will be removed from the scans and replaced by a code and the scans will be saved in a separate archive. The assessor will not have access to the code list.

After the completion of the trial, a blinded assessment of all pseudonymised images will be performed where the investigators assess the images initially assessed by the other investigator. The data will be used to document inter-reader variability.

Additional evaluation of CD activity and disease complication on the MRE and CTE images will be performed using the CDMRIS scale and Lémann Index respectively once all subjects have completed the trial. The CDMRIS scale and Lémann Index are described below. All assessments of the CTE and MRE images will be performed by the investigators at the department of radiology. Only the principal investigator will assess images according to Lémann and CDMRIS.

Other assessments:

During the time the subjects drink the contrast agent prior to the MRE/CTE scan, they will be asked to complete a questionnaire assessing taste, smell, consistency, fullness and ability to swallow the contrast agent.

The subjects will be contacted 2 days after the MRE and CTE examination for control of any potential AE and concomitant medication.

Subjects' experience of anxiety level at the CTE and MRE examinations will be investigated by the use of the State-Trait Anxiety Inventory for Adults questionnaires. The State questionnaire STAI-S consists of 20 statements that evaluate how respondents feel at the moment in terms of tension, apprehension, nervousness, and worry. The inventory might also be used to evaluate how respondents felt at a particular situation in the recent past. STAI-S has been found to be sensitive to changes in transitory anxiety. The Trait questionnaire STAI-T consist of 20 statements that evaluate how respondents feel in general and react to stressful situations. The subjects will respond to the STAI-S directly after the CTE, and MRE, as well as after optional capsule and ultrasound examinations respectively, when remaining at the clinic, and also to the STAI-T directly after the second radiology examination is performed.

A subset of up to 20 subjects will be asked to perform a capsule endoscopy examination and/or ultrasound examination.

* The capsule examination enables visualisation of both the small bowel and the colon mucosa in one procedure. The Crohn's disease severity and presence of strictures, ulcers and other lesions will be evaluated. In the small bowel and colon.
* The ultrasound examination enables visualisation of bowel wall thickening and flow and presence of ulcers, strictures, fistulas and abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender at least 18 years of age at time of signing the informed consent.
* Subjects with a confirmed CD diagnosis
* Clinical indication for an MRE examination of the small bowel, i.e. need for disease status evaluation due to, for example, a relapse/flare, disease status evaluation before starting a new treatment, evaluation of therapeutic effect of given treatment, change in symptomatology, follow-up of longstanding disease, and/or pre-operative mapping/investigation

Exclusion Criteria:

* Clinical suspicion of a severe general or an acute abdominal condition (i.e. bowel obstruction, bowel perforation, severe bleeding or severe inflammation), requiring acute or subacute management.
* Moderate to severe dysphagia
* Known allergy to egg albumin
* Known severe retention of urine
* Known cardiac arrythmia
* Having untreated glaucoma
* Having known manifest thyrotoxicosis
* Having known phenylketonuria
* Having known Glucose-6-phosphatase deficiency
* Contraindicated IV administration of contrast media used in MRE or CTE
* Known sensitivity to any of the components of the investigational product
* Having metallic implants incompatible with MRI examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
RCDAS score | 1 Hour
  Radiological Crohn's Disease Activity Score based on 18 morphologic entities and dynamic signs in the SB and colon. The score range from 0 to 34.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Marsal, Dr., Principal Investigator — Skane University Hospital
Locations (1):
- Department of medical imaging and function, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No